CLINICAL TRIAL: NCT05527470
Title: A Randomized Phase III Prospective Study of Induction Chemotherapy Combined With Concurrent Chemoradiotherapy Versus Induction Chemotherapy Combined With Radiotherapy Alone in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by IMRT or Concurrent Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Lingshan people's Hospital (Unknown); Laibin People's Hospital (Other); Nationalities Hospital of Guangxi Zhuang Autonomous Region (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Principal Investigator, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-08
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Chemoradiotherapy; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Induced Chemotherapy Combined With Radiotherapy Alone in Locoregionally Advanced Nasopharyngeal Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction CT+IMRT Combined Concurrent CT (Active Comparator): Induction Chemotherapy(CT) Followed by Intensity-modulated Radiation Therapy (IMRT ) Combined Concurrent Chemotherapy
  Interventions: Drug: Gemcitabine,Cisplatin; Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin
- Induction CT+IMRT alone (Experimental): Induction Chemotherapy(CT) Followed by Intensity-modulated Radiation Therapy (IMRT )alone
  Interventions: Drug: Gemcitabine,Cisplatin; Radiation: Intensity-modulated radiation therapy (IMRT)

INTERVENTIONS:
Drug: Gemcitabine,Cisplatin — Induction chemotherapy: Patients receive 1000 mg/m2 gemcitabine intravenously on day 1and day 8， 80mg/m2 cisplatin intravenously on day 1 to 3, three cycles were administered at intervals of 3 weeks.
  Other Names: Induction chemotherapy regimen
Radiation: Intensity-modulated radiation therapy (IMRT) — IMRT is given as 2.0-2.3 Gy per fraction with five daily fractions per week for 6-7 weeks, Cumulative doses were > 66 Gy to the primary tumor and > 50 Gy to the bilateral cervical lymph nodes and potential sites of local infiltration.
Drug: Cisplatin — Concurrent chemotherapy: Patients received 100mg/m2 cisplatin intravenously on day 1 to 3, three cycles were administered at intervals of 3 weeks.
  Other Names: Concurrent chemotherapy regimen
  Arms: Induction CT+IMRT Combined Concurrent CT

SUMMARY:
In the era of comprehensive therapy, many studies have investigated the value of induction chemotherapy (IC) in the treatment of nasopharyngeal carcinoma (NPC). Concurrent cisplatin and radiotherapy is the foundation of concurrent chemoradiotherapy strategies, and the addition of cisplatin-based induction chemotherapy to concurrent chemoradiotherapy (CCRT) is considered to prolong survival by reducing distant metastasis in patients with high-risk disease. However, the severity of acute toxicities was significantly increased, which can compromise quality of life and lead to interruptions in CCRT. Fortunately, Locoregional control has substantially improved as the intensity-modulated radiation therapy (IMRT) technique has been widely used in the last decades, IMRT improved the treatment outcomes of patients with NPC, especially the local control rate. Currently, in the era of IMRT, whether patients with NPC benefit from IC plus radiotherapy alone and reduce toxicities compared with IC combined with CCRT. Therefore, the investigators propose this randomized phase III prospective study to assess the efficacy and contribution of IC plus radiotherapy alone in locoregionally advanced NPC during IMRT era.

DETAILED DESCRIPTION:
Patients with stage III-IVA (AJCC 8th, included T1-2N2-3 and/or T3-4N0-3 M0) locoregionally-advanced nasopharyngeal carcinoma will be randomized in a 1:1 ratio to experimental arm and active comparator arm. Patients in experimental arm will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. IMRT is given as 2.0-2.3 Gy per fraction with five daily fractions per week for 6-7 weeks, Cumulative doses were > 66 Gy to the primary tumor and > 50 Gy to the bilateral cervical lymph nodes and potential sites of local infiltration. Patients in active comparator arm will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. IMRT is given as 2.0-2.3 Gy per fraction with five daily fractions per week for 6-7 weeks, Cumulative doses were > 66 Gy to the primary tumor and > 50 Gy to the bilateral cervical lymph nodes and potential sites of local infiltration. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 3 cycles during IMRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type);
2. Tumor staged as III-IVb (according to the 8th AJCC edition);
3. No pregnant female;
4. Age between 18-65;
5. Normal complete blood count level (hemoglobin >10 g/dL, white blood cells ≥4000/μL, platelets ≥100 000/μL);
6. Normal hepatic functions (serum total bilirubin ≤1.6 mg/dL, serum transminase < 2.5 times higher than upper limit);
7. Normal renal function (serum creatinine ≤1.5 mg/dL, creatinine clearance ≥60 mL/min);
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
9. Without radiotherapy or chemotherapy;
10. Patients must give signed informed consent.

Exclusion Criteria:

1. Disease progression in the process of the treatment;
2. The presence of uncontrolled life-threatening illness;
3. History of previous radiotherapy or chemotherapy;
4. Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  Progression-free survival is from randomization to first disease progression [local recurrence and/or distant metastasis] or death from any cause

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Overall survival is from randomization to death of any cause or last follow-up
Locoregional Failure-free Survival | 3 years
  Locoregional failure-free survival is from randomization to locoregional progression
Distant Failure-free Survival | 3 years
  Distant failure-free survival is from randomization to first distant metastasis
Objective response rate | 3 years
  Objective response rate is the percentage of patients achieving complete response (CR) and partial response (PR) according to RECIST 1.1 criteria.
Number of Participants with Adverse Events | 3 years
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi